CLINICAL TRIAL: NCT01557907
Title: Multi-day (3) In-patient Evaluation of Intradermal vs Subcutaneous Basal/Bolus Insulin Infusion
Brief Title: Multi-day (3) In-patient Evaluation of Intradermal Versus Subcutaneous Basal and Bolus Insulin Infusion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BDT-11-ADC001
Record Dates: First submitted 2012-03-09; First posted 2012-03-20 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes
Keywords: Diabetes; Diabetes Mellitus; Type 1 diabetes; Insulin Pump users; Intradermal insulin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal - BD Research Catheter Set (Experimental): Intradermal delivery of insulin (basal and bolus delivery) using the BD Research Catheter Set with 34G x 1.5 mm side-ported needle and the Animas Vibe insulin pump over a three day period.
  Interventions: Device: Intradermal delivery via the BD Research Catheter Set
- Subcutaneous - Medtronic Quick-Set (Active Comparator): Subcutaneous delivery of insulin (basal and bolus delivery) using the Medtronic Quick Set with 6 mm Teflon catheter and the Animas Vibe insulin pump over a three day period.
  Interventions: Device: Subcutaneous delivery via Medtronic Quick-Set

INTERVENTIONS:
Device: Subcutaneous delivery via Medtronic Quick-Set — Infusion rates and pre-meal bolus doses will be based on subjects known daily infusion rate and subject's reported insulin to carbohydrate ratio.
  Other Names: insulin infusion set
  Arms: Subcutaneous - Medtronic Quick-Set
Device: Intradermal delivery via the BD Research Catheter Set — Infusion rates and pre-meal bolus doses will be based on subjects known daily infusion rate and subject's reported insulin to carbohydrate ratio.
  Other Names: microneedles; insulin infusion set
  Arms: Intradermal - BD Research Catheter Set

SUMMARY:
The primary objective of this study is to investigate if intradermal (in the skin) basal and bolus insulin delivery of a fast acting insulin analog (NovoRapid) as needed to adequately control the blood glucose for a subject with Type 1 Diabetes can be maintained for a period of up to three days and if intradermal delivery of insulin has advantages over standard subcutaneous (under the skin) delivery.

DETAILED DESCRIPTION:
The is a single center, open-label, 2 period crossover study randomized by route (intradermal versus subcutaneous) in patients with Type 1 diabetes. Subjects will receive their insulin, basal and bolus dosages, via intradermal (ID) and subcutaneous (SC) infusion sets over a three day period.

Each subject will participate in 3 visits: a Screening Visit (V1), followed by 2 experimental intervention days (V2 and V3) to be started 2 - 21 days after screening visit. The minimum/maximum interval between study days shall be 5 to 28 days. Each subject will remain in the clinic for approximately 3 days during the experimental interventions. A final exam will be performed at the end of Visit 3.

After successful screening and enrollment subjects are admitted to the clinic. Their insulin pump and infusion set is replaced by the investigational system, a commercially available insulin pump and either the intradermal infusion set (Research Catheter Set, BD) or the subcutaneous infusion set (Quick Set, Medtronic)to include an in-line pressure transducer/recorder and insulin NovoRapid. The initial pump infusion rate is established based on the patient's known basal infusion rate and the meal bolus insulin is estimated based on the patient's known insulin sensitivity. An intravenous (in the vein) catheter line is established, blood glucose is measured at least every 2 hours overnight and insulin corrections can be implemented, if deemed necessary. The overnight and pre-prandial (before meal) target range is 70-160 mg/dl, although the procedure will continue as planned if the patient is outside the range. It should be the goal not to give any IV glucose or insulin at all, and not to change basal insulin settings for at least 2 hours before the meal. The breakfast meal will be a high GI (60g carbohydrates) solid meal, to be consumed within 15 minutes and followed for a period of 6 hours of blood sampling for glucose and insulin levels. Lunch will be served as standardized mixed meal, and followed for a period of 4-6 hours. This procedure is repeated on days 2 and 3 whereas the breakfast and lunch meal as well as the insulin dose to cover the meal are the same. A light evening dinner is served every day, composition and insulin dose to be recorded. On day three after the 4 hour period following lunch the catheter will be removed, catheter and site assessments will be documented and an ultrasound observation of the infusion site (skin thickness and SC) versus an adjacent control site will be performed within 10 min after removal of the infusion set. Glucose rescue, if necessary, will be administered orally (juice, 200 mL). Insulin correction boli should be delivered via the investigational infusion set.

ELIGIBILITY:
INCLUSION CRITERIA

Male and Female patients will be included in the trial only if they fulfill all the inclusion criteria mentioned below:

* Understood and signed informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the patient)
* Type 1 Diabetes mellitus, according to clinical judgment / ADA / WHO-definition (Diabetes Care 2003; 26: 5-20) for at least 1 year.
* Usage of insulin pump therapy (CSII) with carb counting for at least six months
* Age in the range of ≥ 18 and ≤ 55 years
* Body mass index (BMI) ≤ 32 kg/m²
* HbA1c ≤ 8.0% at screening
* Using ≤ than 60 U of insulin on a typical day (preferably)
* Able and willing to adhere to the study procedures for the entire trial period
* Negative test results for hepatitis C antibodies, hepatitis B surface antigen and HIV at screening.

EXCLUSION CRITERIA

Patients will not be permitted to enter the trial, if they fulfill any of the exclusion criteria mentioned below:

* Previous participation in this trial or participation in a clinical trial within 3 months prior to screening examination
* Any symptoms suggestive of, or a diagnosis or treatment for gastroparesis
* Abnormalities in renal function (e.g. serum creatinine > 120 µmmol/L for male, >100 µmmol/L for female subjects or judged by the investigator that would pose a problem of clearance of injected insulin
* Proliferative retinopathy or maculopathy that has required acute treatment within the last six months
* Acute and severe illness apart from diabetes mellitus as judged by the investigator
* Abnormalities in the laboratory parameters if judged as clinically significant by the investigator. In particular, patients with GOT/GPT > 3 x upper limit of normal (ULN), thrombocyte count <100/nL, INR >1.3, PTT >50 sec.
* Clinically significant abnormalities in the ECG
* Recurrent major hypoglycemia or hypoglycemic unawareness as judged by the investigator
* Lipodystrophy which in the judgment of the investigator would pose a problem in terms of variability of absorption of injected insulin
* Use of systemic corticoids for the last three month prior screening examination or treatment with medication known to interfere with glucose metabolism such as non-selective ß-blockers, or mono amine oxidase (MAO) inhibitors, ACE-inhibitors or thiazides, unless such medical treatment has existed for at least three months and is not changing, prior to screening examination
* Any disease requiring use of anti-coagulants
* Impaired hepatic or renal functions as judged by the investigator
* Cardiac problems as judged by the investigator
* Uncontrolled hypertension (treated or untreated) RRsyst. >140 mmHg, RRdiast. > 90 mmHg
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Current addiction to alcohol or substances of abuse as determined by the investigator
* Allergy to plaster/adhesive
* Any other condition that the investigator feels would interfere with trial participation or evaluation of results.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Insulin levels | 0,10,15,20,25,30,35,40,45,50,55,60,65,70,80,90,120,150,180,210,240,300,330,345,360 minutes following each breakfast and lunch meal bolus for the 3 study days
  Time to peak plasma concentration (Tmax) of insulin delivered intradermally as compared to insulin delivered subcutaneously after a meal bolus.

SECONDARY OUTCOMES:
Insulin levels | 0,10,15,20,25,30,35,40,45,50,55,60,65,70,80,90,120,150,180,210,240,300,330,345,360 minutes following each breakfast and lunch meal bolus for the 3 study days
  Comparison of peak plasma concentration (Cmax) of insulin, intradermally versus subcutaneously, during a meal bolus period.
  Comparison of area under the plasma concentration versus time curve (AUC), intradermally versus subcutanously, during a meal bolus period.
Blood Glucose | 0,10,15,20,25,30,35,40,45,50,55,60,65,70,80,90,120,150,180,210,240,300,330,345,360 minutes following each breakfast and lunch meal bolus for the 3 study days
  Peak concentration of blood glucose (BGmax) during post meal excursions periods.
  Area under the plasma concentration versus time curve (AUC) of blood glucose during post meal excurion periods.
Device performance - adhesion | Evaluated at every timepoint a bolus injection is given
  Adhesion (device remains attached to the skin) will be evaluated over the 3 day study period (adhered well, partially adhered, completely pulled off).
Skin thickness using ultrasound | Upon removal of the device (within 5 minutes)
  Skin thickness will be measured at the infusion site and a control site using ultrasound
Device performance - Leakage of fluid (insulin) at injection site | Immediatley before and after each bolus injection and immediatly upon removal of the device at the end of the study period.
  Immediatley before and after each bolus injection, the site will be observed for leakage (insulin). In addition, following removal of the device, if leakakge is observed, the fluid will be collected and quantified using a gravimetic method procedure. Leakage will be collected using a pre-weighed sterile absorbent swab, the swab will be re-weighed and the collected fuid volume calculated based on the density of the fluid.
Device performance-pump alarm | over the 3 study days
  The presence of an auditory alarm indicating an occlusion will be noted.
Skin effects-Draize Scoring for Skin Irritation | Following removal of the device (within 2 minutes) and 1 and 2 hours (+/- 5 minutes) post removal.
  Local reaction at injection site will be scored using the Draize Scale 0-4 for redness and 0-4 for swelling.
Number of participants with adverse events | up to 53 days or until the subject is discharged, if sooner.
  At each study contact, subjects will be questioned about any new or worsening undesirable events.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, MD, Principal Investigator — Profil Institut fur Stoffwechselforschung (GmbH)
Locations (1):
- Profil Institut fur Stoffwechselfforschung GmbH, Neuss, Germany